CLINICAL TRIAL: NCT01826877
Title: A Phase I, Open Label, Dose Escalation and Cohort Expansion Study to Evaluate the Safety and Immune Response to Autologous Dendritic Cells Transduced With Ad-GMCAIX in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Autologous Dendritic Cells in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Kite, A Gilead Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-000577; NCI-2013-00646 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-04; First posted 2013-04-09 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (autologous dendritic cells) (Experimental): Patients receive AdGMCAIX-transduced autologous dendritic cells ID on days 1, 15, and 29.
  Interventions: Biological: AdGMCAIX-transduced autologous dendritic cells; Biological: therapeutic autologous dendritic cells; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: AdGMCAIX-transduced autologous dendritic cells — Given ID
  Other Names: DC-AdGMCAIX; dendritic cells transduced with AdGMCA9 expressing GM-CSF-carbonic anhydrase IX fusion protein
Biological: therapeutic autologous dendritic cells — Given ID
  Other Names: ADC; autologous dendritic cells
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of autologous dendritic cells in treating patients with metastatic kidney cancer. Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of dendritic cell (DC)-AdGM carbonic anhydrase IX (CAIX) administered by intradermal injections at study doses and schedule.

SECONDARY OBJECTIVES:

I. To evaluate clinical antitumor effects following study treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1. Parameters include objective response (complete response [CR], partial response [PR]), duration of response in patients with objective response, and time to disease progression.

II. To evaluate immune responses to DC-AdGMCAIX vaccination by enzyme-linked immunospot (ELISpot) for numeric determination of CAIX specific T cells in blood.

III. To evaluate immune responses to DC-AdGMCAIX vaccination by cytokine profiling of T cell culture supernatants for characterization of the immune response in subjects with demonstrated immune activation may be performed.

IV. To evaluate immune responses to DC-AdGMCAIX vaccination by anti-sargramostim (GM-CSF) antibody response.

V. To evaluate tumor biopsies for immune cell infiltrates.

OUTLINE: This is a dose-escalation study.

Patients receive AdGMCAIX-transduced autologous dendritic cells intradermally (ID) on days 1, 15, and 29.

After completion of study treatment, patients are followed up every 2-3 months for at least 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed clear cell renal cell carcinoma (ccRCC); pathology report from the original diagnosis of renal cell carcinoma is acceptable; the component of conventional clear cell type > 50% is mandatory
* Evidence of metastatic disease with measurable lesion(s) as defined by RECIST guideline version 1.1 to permit tumor response evaluation; subjects with unresected primary tumors may be enrolled as long as evidence of measurable metastatic disease is also present
* Signed informed consent
* Eastern Cooperative Oncology Group (ECOG) =< 1
* Expected life expectancy >= 6 months
* Serum creatinine < 2 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 X upper limit of normal (ULN)
* Total bilirubin < 2 X ULN (except for subjects with documented Gilbert's syndrome who can have total bilirubin < 3.0 mg/dl)
* Hemoglobin >= 10 g/dL
* Absolute neutrophil count >= 1.5 X 10^9 cells/L
* Platelets >= 100 X 10^9/L
* Having recovered from prior surgery, radiation, chemotherapy (cytotoxic and noncytotoxic) to toxicity grade =< 1 or returned to baseline; previous treatment with immunotherapies, cytotoxic drugs, or other targeted agents is permitted; if cytotoxic chemotherapy was previously received, the last dose must be >= 1 month before leukapheresis; for other agents, the last dose must be >= 14 days before leukapheresis
* Negative serum pregnancy test within 7 days prior to enrollment in female subjects with reproductive potential

Exclusion Criteria:

* Rapidly progressing cancer likely to require palliative systemic intervention within 8 weeks after study entry
* Presence of untreated/active central nervous system (CNS) metastases
* For subjects with metastatic RCC who have had no prior systemic treatment for RCC and are considered a poor risk according to Motzer criteria, defined by having >= 3 of the following 5 risk factors for short survival: Karnofsky performance score < 80%, lactate dehydrogenase (LDH) > 1.5 X of ULN, hemoglobin < lower limit of normal (LLN), corrected serum calcium > 10 mg/dL (2.5mM), a time from initial diagnosis of RCC to initiation of systemic therapy of < 1 year
* Non-clear cell or predominantly (> 50%) sarcomatoid histology
* Concurrent major medical conditions, such as uncontrolled hypertension, diabetes mellitus, ischemic heart disease, chronic obstructive pulmonary disease, autoimmune disease, adrenal insufficiency, or prior allogeneic organ transplant requiring chronic immunosuppressive therapy, including systemic glucocorticoid treatment or replacement therapy
* Active or chronic systemic infection, including viral hepatitis, human immunodeficiency virus (HIV), mycobacteria, tuberculosis (TB), or other opportunistic infections
* Having received systemic immune suppressive therapy within 30 days prior to leukapheresis
* Having received an investigational agent within 30 days prior to the first dose of study treatment
* Female subjects who are lactating, pregnant or both male and female subjects with reproductive potential who refuse to practice medically accepted methods for contraception over the period from study consent to 90 days following the last dose of study treatment
* Other malignancy within 3 years, except for adequately treated non-melanoma skin cancer, non-invasive cancers such as cervical or breast carcinoma in situ, or superficial bladder cancer without local recurrence
* Social or psychological conditions that the investigator judges may compromise study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events including all grade 3 and grade 4 adverse events regardless of causality, treatment-related adverse events, dose limiting toxicities (DLT), and adverse events leading to discontinuation of study treatment | Up to day 57
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03

SECONDARY OUTCOMES:
CAIX-specific immune response | Up to 3 years
  Measured by ELISpot analysis of T cells from blood and cytokine profiling in T cell cultural supernatants.
Objective response (CR, PR) according to RECIST guideline version 1.1 | Up to 3 years
Duration of progression-free survival | Up to 3 years
Clinical benefit rate (CR, PR, and SD) greater than or equal to 12 weeks | Up to 3 years
Disease response (CR, PR, stable disease [SD], and progressive disease [PD]) according to RECIST guideline version 1 | Up to 3 years
Duration of response according to RECIST guideline version 1 | Up to 3 years
Time to disease progression | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Drakaki, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Faiena I, Comin-Anduix B, Berent-Maoz B, Bot A, Zomorodian N, Sachdeva A, Said J, Cheung-Lau G, Pang J, Macabali M, Chodon T, Wang X, Cabrera P, Kaplan-Lefko P, Chamie K, Belldegrun AS, Pantuck AJ, Drakaki A. A Phase I, Open-label, Dose-escalation, and Cohort Expansion Study to Evaluate the Safety and Immune Response to Autologous Dendritic Cells Transduced With AdGMCA9 (DC-AdGMCAIX) in Patients With Metastatic Renal Cell Carcinoma. J Immunother. 2020 Nov/Dec;43(9):273-282. doi: 10.1097/CJI.0000000000000336. PMID 32925563